CLINICAL TRIAL: NCT03152357
Title: A Retrospective Study to Evaluate the ConforMIS iUni, iDuo & iTotal® CR (Cruciate Retaining) Knee Replacement Systems
Brief Title: A Retrospective Study to Evaluate the ConforMIS iUni, iDuo & iTotal® KRS
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-003
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee; Knee Osteoarthritis
Keywords: osteoarthritis; total knee arthroplasty; TKA; TKR; patient specific; Conformis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients implanted with a ConforMIS device: Previously underwent surgical implantation of a ConforMIS iUni, iDuo or iTotal knee replacement
  Interventions: Device: ConforMIS iUni, iDuo, or iTotal (CR)

INTERVENTIONS:
Device: ConforMIS iUni, iDuo, or iTotal (CR) — ConforMIS iUni, iDuo, or iTotal (CR)

SUMMARY:
This study is designed to evaluate implant survivorship, patient satisfaction, and patient-reported outcomes of subjects who have undergone surgery with any of the following ConforMIS knee implants: the iUni®, iDuo® or iTotal® Cruciate Retaining (CR) Knee Replacement Systems.

DETAILED DESCRIPTION:
This study is designed to evaluate implant survivorship, patient satisfaction and patient-reported outcomes of subjects who have undergone surgery with any of the following ConforMIS knee implants: the iUni®, iDuo® or iTotal® Cruciate Retaining (CR) Knee Replacement Systems.This study is a retrospective, single-center study, with one single remote follow up contact. Patients will be contacted either by phone or email for a single remote follow-up. Retrospective data will be collected from medical records including pre-operative, operative and any follow up visits which have occurred since implantation as available.

ELIGIBILITY:
Inclusion Criteria:

* Previously underwent surgical implantation of a ConforMIS iUni, iDuo or iTotal knee replacement.
* Subject must be greater than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's over 18 that have undergone surgical implantation of a ConforMIS product
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Survivorship data | 1 year
  Survivorship of the implant--whether or not the patient has had a surgical revision prior to data collection.

SECONDARY OUTCOMES:
Patient Reported Outcomes | 1 year
  Collected via questionnaires during either an in-office visit or a phone call. The questionnaires are aimed at gauging how satisfied the patient is with the function of their device, if and when they experience pain/stiffness, and if and how their activities of daily living have have been affected.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Martin, MD, Principal Investigator — JFK Medical Center
Locations (1):
- Preferred Orthopedics of the Palm Beaches, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Fitzpatrick C, FitzPatrick D, Lee J, Auger D. Statistical design of unicompartmental tibial implants and comparison with current devices. Knee. 2007 Mar;14(2):138-44. doi: 10.1016/j.knee.2006.11.005. Epub 2006 Dec 22. PMID 17188876
- [Background] Fitz W. Unicompartmental knee arthroplasty with use of novel patient-specific resurfacing implants and personalized jigs. J Bone Joint Surg Am. 2009 Feb;91 Suppl 1:69-76. doi: 10.2106/JBJS.H.01448. PMID 19182028
- [Background] Rougraff BT, Heck DA, Gibson AE. A comparison of tricompartmental and unicompartmental arthroplasty for the treatment of gonarthrosis. Clin Orthop Relat Res. 1991 Dec;(273):157-64. PMID 1959265
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035